CLINICAL TRIAL: NCT02469285
Title: The Effect of Pork With Modified Fatty Acid Composition on Plasma Lipids and Fatty Acids and the Effect of Pork and Berries on Fecal Compounds in Healthy Adults
Brief Title: The Effect of Pork With Modified Fat Composition and Berries on Plasma Fatty Acids and Fecal Compounds in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Anne-Maria Pajari, Adjunct professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KarniMari-HY
Record Dates: First submitted 2014-12-21; First posted 2015-06-11 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases
Keywords: Fatty acids; Lipids; Nitroso compounds; Lipid metabolism; Gut metabolism
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Pork Meat; Fruit

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Modified pork (Experimental): Pork with modified fatty acid composition, more unsaturated fat. 160 g pork or pork products daily for 4 weeks, consumption of other red meat is prohibited
  Interventions: Dietary Supplement: Modified pork
- Normal pork (Active Comparator): Normal pork 160 g pork or pork products daily for 4 weeks, consumption of other red meat is prohibited
  Interventions: Dietary Supplement: Pork
- Normal pork and berries (Experimental): Normal pork and berries (strawberry, raspberry, wild blueberry, lingonberry, cloudberry, blackcurrant) 160 g pork or pork products daily for 4 weeks, consumption of other red meat is prohibited
  Interventions: Dietary Supplement: Pork and berries

INTERVENTIONS:
Dietary Supplement: Modified pork — Pork with modified fatty acid composition
  Other Names: Pork with modified fatty acid composition and berries; Pork; Pork and Finnish berries
  Arms: Modified pork
Dietary Supplement: Pork — Pork with normal fat composition
  Arms: Normal pork
Dietary Supplement: Pork and berries — Pork with normal fat composition and Finnish berries
  Arms: Normal pork and berries

SUMMARY:
High consumption of red meat is related to cardiovascular diseases. Red meat containing more unsaturated fat than normal red meat may have a beneficial impact on plasma lipid and fatty acid profile in humans. Furthermore, consumption of red meat and especially processed red meat is considered harmful to colon health. However, consumption of fruit and berries rich in antioxidants and flavonoids may provide protection when red meat is consumed.

The study aims to answer whether the fatty acid profile of pork when modified towards more unsaturated fat will affect plasma fatty acids and lipids in adult volunteers. The effects of pork with a modified fatty acid content is compared with conventional pork with lower unsaturated fat content. Fatty acid composition of pork is modified by altering the composition of animal feed.

The other arm of the study investigates the effects of consuming berries together with red meat on gut metabolism. The study focuses on how berries affect the formation of fecal compounds known to be related to high red meat consumption, such as N-nitroso compounds.

ELIGIBILITY:
Inclusion Criteria:

* diet includes meat

Exclusion Criteria:

* high consumption of fish (4 times per week)
* use of fish oil/ omega-3 oil capsules one month before the intervention
* hypercholesterolemia
* vegetarian, vegan

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in plasma fatty acids as a measure of dietary fatty acid modification | 4 weeks
Change in fecal nitroso compounds as a measure of increased (processed) red meat consumption | 4 weeks
  Measured as apparent total nitroso compounds (ATNC)
Genotoxicity testing of human fecal water in 3D cell culture | 4 weeks
  Fecal water is isolated from fecal samples collected before and after the intervention period from arms B and C. The samples are tested for markers of genotoxicity in 3D cell culture.

SECONDARY OUTCOMES:
Changes in plasma lipids as a measure of dietary modification | 4 weeks
  Concentrations of and changes in total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides are measured before and after the intervention period
Concentration of polyphenolics in fecal water as a measure of consumption of berries | 4 weeks
  The polyphenol content of the fecal water is assessed from arms B and C
Change in hemoglobin as a measure of dietary modification | 4 weeks
Change in blood pressure as a measure of dietary modofcation | 4 weeks
  Blood pressure is measured before and after the study period.
Weight development during the study period | 4 weeks
  The subjects are weighed before and after the study and their weight is monitored weekly during the study

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maria Pajari, PhD, Principal Investigator — Division of Nutrition, Department of Food and Environmental Sciences, University of Helsinki; Marja Mutanen, PhD, Principal Investigator — Division of Nutrition, Department of Food and Environmental Sciences, University of Helsinki
Locations (1):
- Division of Nutrition, University of Helsinki, Helsinki, Finland